CLINICAL TRIAL: NCT02538237
Title: A Randomized, Double-Blind, Split-mouth, Placebo-controlled, Clinical Trial of the Effect of Sub-gingival Irrigation With Ibuprofen Mouthwash in Treatment of Periodontal Diseases
Brief Title: the Effect of Sub-gingival Irrigation With Ibuprofen 2% Mouthwash in Treatment of Periodontal Diseases.
Acronym: ibuprofen
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Amirhossein Farahmand, assistant prof, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: subgingival irrigation
Record Dates: First submitted 2015-08-29; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Ibuprofen; Mouthwashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ibuprofen mouthwash (Experimental): Subgingival Irrigation of ibuprofen 2% mouthwash (made from the Faculty of Pharmaceutical Sciences, Islamic Azad University, Tehran) with an insulin syringe 0.5 ml were rinsed
  Interventions: Drug: Ibuprofen 2% mouthwash
- placebo mouthwash (Sham Comparator): Subgingival Irrigation of placebo 2% mouthwash (made from the Faculty of Pharmaceutical Sciences, Islamic Azad University, Tehran) with an insulin syringe 0.5 ml were rinsed
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — the mouthwash(ibuprofen 2% or placebo) Subgingival Irrigation of mouthwash with an insulin syringe 0.5 ml were rinsed.
  Other Names: Ibuprofen 2% mouthwash (made from the Faculty of Pharmaceutical Sciences, Islamic Azad University, Tehran)
  Arms: placebo mouthwash
Drug: Ibuprofen 2% mouthwash
  Arms: ibuprofen mouthwash

SUMMARY:
Aim: Use an ibuprofen mouthwash 2% irrigate subgingival in improving the progression of periodontal diseases can be evaluated. Materials and Methods: 22 patients with chronic periodontitis without any systemic disease who have had periodontal disease, and 2 molars that have periodontal pockets deeper than 4 mm on either side of the lower jaw have the clinical examinations. Interventions: For patients who participated in this study, subjects who received oral hygiene instruction and scaling root planing (SRP), After 2 weeks, They were divided into two groups as determined by randomization in this study, Experimental group: ibuprofen 2% mouthwash (made from the Faculty of Pharmaceutical Sciences, Islamic Azad University, Tehran), Control group: placebo, Subgingival Irrigation of ibuprofen 2% mouthwash with an insulin syringe 0.5 ml were rinsed, Clinical measurements including probing depth (PD), clinical attachment levels (CAL), Plaque Index (PI), and Bleeding Index (BI) were recorded and the patients were recalled per once every 2 weeks for 3 months is repetitive, and at the end of 3 months, were evaluated changes in clinical periodontal parameters. ®

DETAILED DESCRIPTION:
Patients and methods

Eligible participants were 22 adult patients treated for chronic periodontitis and participating in a supportive periodontal therapy program at the Department of Periodontology of the Dental Clinic of the Islamic Azad University, Dental Branch of Tehran were included in the current study; Recruitment of participants started November 2013 and ended September 2014. The study met the criteria of the Helsinki Declaration of1975, revised in 2008. The survey plan was reviewed and sanctioned, approved by the ethics commission of the Institutional Ethical Committee and Review Board of the Deputy of Research, School of Dentistry. All subjects received the oral and written explanation of the intent of the survey and signed an informed consent after receiving detailed information about the purpose, the benefits, and the possible risks associated with the trial. Individuals satisfying the following entry criteria were recruited:

* Diagnosed suffering from initial (early) to moderate chronic periodontitis;
* Adult patients, more than 28 years old with at least 20 remaining teeth and at least three teeth in each quadrant;
* The presence of at least two residual sites with a probing pocket depth (PPD≥4 mm in two opposite quadrants, which showed bleeding upon probing, radiographically comparable amount of periodontal breakdown and good matching in tooth type, also clinical and minimal radiographic signs of initial (early) to moderate (clinical attachment level of 1 to 3mm.

Exclusion criteria:

Periodontal treatment (non-surgical) the previous six months Systemic diseases; Hypersensitive to Ibuprofen; Systemic antibiotic or anti-inflammatory drugs within the three months preceding the beginning of the study; Pregnant or nursing females; Smoking; No acute periodontal conditions, such as necrotizing periodontal diseases or periodontal abscesses. Mouth rinses during the entire period of the study orthodontic treatments, Use of removable dentures, Extensive dental restorations.

Clinical measurements

The following clinical outcome variables were recorded at baseline, within 7 days to 3 months at the selected teeth, at six sites per tooth, by means of a periodontal probe (William's® probe, Hu-Friedy, USA) by two calibrated blinded examiners:

* Plaque index (PI) using a Silness & Loe index (18).
* Bleeding on probing (BOP), through the visual inspection 30 s after probing, (Score 0: No bleeding after probing. Score 1: A single discrete bleeding point appears after probing) (19).
* Probing pocket depth (PPD) in millimeters, measured from the gingival margin to the deepest stop of the periodontal pocket at the standardized force.
* Clinical attachment level (CAL), calculated by adding PPD at each site.

Examiner calibration and reproducibility were ensured by duplicating measurements of four periodontitis patients, not included in the study, with a one-day interval, prior to the start of the survey. Repetitive measurements were within a 1mm difference in 91.5 % of the recordings.

Study design and interventions the study was a randomized, placebo-controlled, parallel, split-mouth designed 3-months clinical trial.

Treatment phase I: instruction on oral hygiene procedures after having entered the study, all patients received the following procedures:

* Individualized oral hygiene instructions together with the provision of a new toothbrush, dental floss, and a fluoridated dentifrice.
* Full-mouth periodontal examination ultrasonic instruments and supragingival professional prophylaxis using.

Treatment phase II: After patient selection; using blocked randomization with a block size of 4 and an allocation ratio of 1:1 Block randomization was chosen to prevent too much variability in the number of patients randomized and ensure a reasonably steady flow of patients to each treatment group, Allocation cover was ensured by using container and labeling that did not reveal the content of the trial drug packages who was blind to the therapist and the clinical examiner. Also, the test and placebo mouthwashes had a similar color. Patients were randomly assigned to either the A or B group, while mandibular arches are each divided into two parts (left and right sections);about 60 sites in both groups; individuals received scaling and root planing on the first visit in accordance with the one-stage full-mouth debridement protocol (scaled by means of an ultrasonic device) + professional cleaning; The therapeutic endpoint was defined as a clean root surface without visible or clinically detectable remnants of biofilm or calculus, since two weeks, the mouthwashes were applied into the periodontal pockets with PD ≥4 mm using a syringe with a blunt cannula; and After isolating and drying the selected sites, the assigned ibuprofen mouthwash 2% formulation (made by Islamic Azad university pharmaceutical sciences branch) was subgingivally applied using a needle with a blunt tip and a lateral opening for avoiding any trauma to the tissues. Follow-up visits were scheduled after 0, 7, 14 days, within three months. At these visits, the following clinical outcome variables were recorded at baseline and within seven days to three months at the selected teeth by William's periodontal probe; at six sites per tooth. Oral hygiene was reinforced at each visit, but no further treatment was provided. Within any visit, patients were provided with a full-mouth professional prophylaxis. At every visit, the occurrence of any undesirable side effects or adverse events that could be related to the treatment was recorded, including changing of both teeth and oral mucosa.

Statistical analyses the sample size is calculated using the following formula: α=00.05 and the power (1-β) =80%. For the variability (σ = SD), the value of 0.5 mm was used, considering PPD change from baseline to three months as the main outcome variable, with a desired difference of 1.8 mm. On the basis of these data, the number of enrolled patients to conduct this study was calculated as 12 patients per arm. However, considering the possibility of having a certain amount of drop outpatients (10%), the total number of requests patients was 14 per treatment group. Statistical methods only the data from the selected sites were processed, but the patient was considered the statistical unit. The obtained clinical outcome variables were calculated by the patient, and then by treatment group. For the evaluation of the intragroup changes between baseline and 7, 14, within three months the ANOVA test was used (once the normality of the distribution was proven). Statistical significance was defined as P <0.001. All data were analyzed using a software program (SPSS 19).

ELIGIBILITY:
Inclusion Criteria:

* The patients systemically healthy were selected for the study.
* The subjects had with periodontal pocket depths of more than 4 mm on at least two teeth in the mandibular molar area that observed on probing.

Exclusion Criteria:

* Existing systemic disease;
* Hypersensitive to Ibuprofen;
* The use of any Antibiotic or Anti-inflammatory drugs within the 6 months preceding the beginning of the study;
* Cancer;
* Pregnant or nursing females;
* Smoking; Orthodontic treatments;
* Extensive dental restorations;
* Use removal denture;
* Mouth rinses;
* during the entire period of the study.

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Reduction of periodontal pocket | 15 days
  periodontal probe

SECONDARY OUTCOMES:
Reduction of bleeding on probing | 3 months
  periodontal probe